CLINICAL TRIAL: NCT04971967
Title: Enhancing Partner Services Among Men Who Have Sex With Men Living With HIV: A Pilot Randomized Controlled Trial
Brief Title: Enhancing Partner Services Among Men Who Have Sex With Men Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-0496; R34MH119963 (NIH)
Record Dates: First submitted 2021-06-29; First posted 2021-07-22 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-09

CONDITIONS: Contact Tracing
Keywords: Partner notification services; Crowdsourcing; MSM; HIV

STUDY DESIGN:
Intervention Model Description: 120 newly identified MSM HIV cases will be randomly assigned into two groups in 2:1 ratio (intervention: control) and receive crowdsourced PS and conventional PS, respectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crowdsourced HIV PS Group (Experimental): Participants in the intervention group will receive crowdsourced partner services intervention, including postcards from the crowdsourcing contest that promote PS, provider referral and dual referral services, and take-home HIV self testing kits.
  Interventions: Combination Product: Crowdsourced partner services intervention
- Conventional HIV PS Group (No Intervention): Participants in the control group will receive traditional partner services intervention, including referral cards that encourage the index patient to notify their partners by themselves.

INTERVENTIONS:
Combination Product: Crowdsourced partner services intervention — The intervention includes the provision of provider referral and dual referral services, crowdsourced materials such as postcards and an HTML aiming to promote PS, as well as free take-home HIV self-testing kits.
  Arms: Crowdsourced HIV PS Group

SUMMARY:
Individuals will participate in a pilot randomized controlled trial (RCT) that implements and evaluates the feasibility, acceptability, and effectiveness of crowdsourced partner services (PS) or conventional PS among Chinese men who have sex with men (MSM) living with HIV.

The pilot RCT will include 120 newly identified MSM HIV cases who were born biologically male, aged 18 years old or older, newly identified as HIV positive, had oral or anal sex with a man, had at least one sexual partner in the previous 6 months and live in Guangzhou. Participants will undergo a series of computer-based interviews (baseline and 2 months after enrollment) and will be randomly assigned into two groups in 2:1 ratio (intervention: control) and receive crowdsourced PS and conventional PS, respectively.

DETAILED DESCRIPTION:
This is a pilot RCT, and the primary outcomes of this study are: 1) to test the feasibility and acceptability of the crowdsourced intervention, and 2) to pilot the preliminary impact of crowdsourced PS intervention in promoting HIV testing among partners of the newly identified HIV cases. In addition, this pilot RCT aimed to collect preliminary data for the designing of a full RCT, which aimed to measure the efficacy of the crowdsourced PS intervention in promoting PS. Thus, the sample size of this study is not designed and will be not powered enough to test the difference between the two arms. However, with a sample size of 120 (80 for intervention arm and 40 for the control arm, respectively), this pilot study would be able to observe the differences between the two arms and collect preliminary data for adequate sample size calculation of a full RCT. With a sample size of 120 (ratio of 2:1), alpha=0.05, power=0.80, and the partner return rate in the conventional PS arm is 30% (around 31% in 2016 in Guangzhou), the minimal detectable effect size would be 26.7% for this pilot study.

Data analyses: For the primary outcomes of feasibility and acceptability of the intervention: this will be analyzed through descriptive analysis to assess the feedback on the feasibility and acceptability of the crowdsourced PS intervention at baseline and the follow-up survey. For the primary outcome of the proportion of partners returning for HIV testing within 2 months of the index participant's enrolment in the study, log-binomial regression (generalized linear model with binomial distribution and log link) will be used to calculate 95% confidence intervals for the proportion of notifiable partners visiting by arm. Risk differences and risk ratios will also be calculated in these models. As this study is a pilot RCT, adjustment for covariates is not necessary and will not be conducted in the primary analysis. In secondary analyses, pre-specified potential confounding variables will be adjusted that might bias the estimate if not accounted for (e.g. index age, index marital status). If a partner reports more than one index referred him, he will be counted as a returning partner for each identified index.

Subgroup analyses will be performed by partner sex, partner type (e.g. main male partner vs. casual male partner) and sexual orientation. Time to presentation will also be assessed among all notifiable partners using Cox proportional hazards with a robust variance estimator. In the time-to-event analyses, censoring will occur at the end of 2-months. Note that for the primary outcome, the assumption is that any partner without an identifiable record at the community center or in the centralized electronic medical record (EMR) did not present for HIV testing. Therefore, this study assumes no missing outcome data. Sensitivity analyses will be conducted using alternative definitions of presentation for testing, including using the self-reported data from index cases and partners. For count variables expressed as the mean number of partners, the investigators will use either Poisson regression or negative binomial regression if overdispersion is identified.

ELIGIBILITY:
Inclusion Criteria:

* born biologically male,
* aged 18 years old or older,
* newly identified as HIV positive,
* had oral or anal sex with a man,
* had at least one sexual partner in the previous 6 months
* live in Guangzhou

Exclusion Criteria:

* Not meet inclusion criteria
* Not given informed consent

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Tang, Ph.D, Principal Investigator — University of North Carolina Project-China
Locations (1):
- Guangzhou Center for Diseases Control and Prevention, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: The investigator who proposes to use the data needs to have approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Yan X, Tucker JD, Miller WC, Xu H, Zhou Y, Gu Y, Chen M, Liang M, Lu J, Zhan L, Tang W. Crowdsourced Partner Services Among Men Who Have Sex With Men Living With HIV: A Pilot Randomized Controlled Trial in China. Sex Transm Dis. 2024 Oct 1;51(10):673-680. doi: 10.1097/OLQ.0000000000001989. Epub 2024 May 1. PMID 38691408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three HIV testing clinics were selected as recruitment sites; they were based at Guangzhou CDC, an MSM CBO in Guangzhou, and an MSM CBO in Zhuhai, respectively. The baseline recruitment lasted from August 1st 2021 to May 26th 2022.
Groups:
- Crowdsourced HIV PS Group: Participants in the intervention group will receive crowdsourced HIV partner services that integrated three parts: (a) educational materials for HIV PS promotion purposes, (b) secondary distribution of HIVST kits (HIVST-SD) to sexual partners, and (c) options of provider referral or contract referral using anonymous notification messages.
  The educational materials included (a.1) postcards from previous crowdsourcing events to facilitate HIV PS, and (a.2) a digital platform embedded in the WeChat application that offered HIV PS skills by partner types, and potential risks or adverse consequences. The digital platform also included a section on peer sharing, where MLWH shared their experience of successfully disclosing their HIV status to their sexual partners in text or video forms. The QR code of the digital platform was printed on (a.3) a public transport card pre-charged with $3 for portable usage and easy access.
- Conventional HIV PS Group: Participants in the control group will receive traditional partner services intervention, which uses referral cards that encourage the index patient to notify their partners by themselves.
Period: Overall Study
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Started | 81 | 40
Completed | 75 | 33
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group | Total
Number analyzed (Participants) | 81 | 40 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.1) | 31.0 (9.6) | 30.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 81 | 40 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 81 | 40 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 81 | 40 | 121
Sexual orientation [Count of Participants; unit: Participants]
  Gay | 56 | 35 | 91
  Straight | 4 | 2 | 6
  Bisexual | 18 | 3 | 21
  Other/Prefer not to answer | 3 | 0 | 3
Sexual orientation disclosure [Count of Participants; unit: Participants]
  Yes | 64 | 31 | 95
  No | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of MSM Index Cases That Respond to the Follow-up Survey at 3 Months After Enrollment
Description: Intervention feasibility, measured by the percentage of MSM index cases that respond to the follow-up survey 3 months after enrollment
Time Frame: 3 months post enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 81 | 40
percentage of participants | 92.6 [84.8 to 96.6] | 82.5 [68.1 to 91.3]

2. Primary Outcome: Acceptability Degree of the Intervention Using an Acceptability Questionnaire
Description: Intervention acceptability, measured by the mean score of an acceptability questionnaire among index patients in the intervention group at 3-month follow-up. The questionnaire asks index patients about their responses to statements regarding the acceptability of the crowdsourced intervention materials, and is rated on a 1-5 scale with mean scores ranging between 1 and 5, where 1 means 'strongly disagree' and 5 means 'strongly agree'. Higher mean scores mean higher acceptability.
Time Frame: 3 months post enrollment
Population: Only indexes in the intervention arm who completed the 3-month follow-up survey would provide acceptability data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 75 | 0
score on a scale | 4.4 (1.1) |

3. Primary Outcome: Percentage of Partners Who Perform HIV-testing Within 3 Months of the Index Patient's Enrollment
Description: The preliminary impact of the intervention, measured by the percentage of partners who perform HIV-testing within 3 months of the index patient's enrollment. Partner HIV testing is self-reported by the index, and verified by the partners uploading testing results.
Time Frame: 3 months post enrollment
Population: 81 indexes in the intervention arm reported 171 sexual partners in total, and 40 indexes in the control arm reported 89 sexual partners in total.
Measure: Number (95% Confidence Interval); unit: percentage of partners
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 171 | 89
percentage of partners | 38.0 [31.1 to 45.5] | 27.0 [18.8 to 37.0]
Statistical Analysis 1: Comparison: Crowdsourced HIV PS Group vs Conventional HIV PS Group; Test type: Superiority; p = 0.07, Generalized linear regression

4. Secondary Outcome: Percentage of Partners Who Were Notified Within 3 Months of the Index's Enrollment
Description: The percentage of partners who were notified by their indexes within 3 months of the index's enrollment
Time Frame: 3 months post enrollment
Population: 81 indexes in the intervention arm reported 171 sexual partners, and 40 indexes in the control arm reported 89 sexual partners.
Measure: Number (95% Confidence Interval); unit: percentage of partners
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 171 | 89
percentage of partners | 34.5 [27.8 to 41.9] | 28.1 [19.8 to 38.2]
Statistical Analysis 1: Comparison: Crowdsourced HIV PS Group vs Conventional HIV PS Group; Test type: Superiority; p = 0.30, Generalized linear regression

5. Secondary Outcome: Mean Number of Partners Tested Per Index
Description: The mean number of sexual partners tested per index followed for the last 3 months.
Time Frame: 3 months post enrollment
Population: Only index participants who finished the 3-month follow-up survey were included for analysis, including 75 out of 81 participants in the intervention group, and 33 out of 40 participants in the control group.
Measure: Mean (Standard Deviation); unit: tested partners per index
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 75 | 33
tested partners per index | 0.9 (1.3) | 0.7 (0.7)

6. Secondary Outcome: Percentage of Partners Who Have Positive HIV Tests Among All Tested Partners
Description: The percentage of partners tested as HIV positive among partners who performed HIV-testing in the last 3 months.
Time Frame: 3 months post enrollment
Population: 65 sexual partners received HIV testing in the intervention group, and 24 sexual partners received HIV testing in the control group.
Measure: Number (95% Confidence Interval); unit: percentage of partners
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 65 | 24
percentage of partners | 23.1 [14.5 to 34.6] | 12.5 [4.3 to 31.0]
Statistical Analysis 1: Comparison: Crowdsourced HIV PS Group vs Conventional HIV PS Group; Test type: Superiority; p = 0.28, Generalized linear regression

7. Secondary Outcome: Mean Number of Case-finding Per Index
Description: The mean number of case-finding (i.e., partners tested positive) per index within 3 months post index enrollment
Time Frame: 3 months post enrollment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: positive partners per index
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 75 | 33
positive partners per index | 0.2 (0.4) | 0.1 (0.4)

8. Secondary Outcome: Percentage of Casual Male Partners Getting HIV Testing
Description: The percentage of partners getting HIV testing who are not spouses or regular male partners
Time Frame: 3 months post enrollment
Population: Only casual male partners reported by index participants were included in this analysis, including 110 casual male partners from the intervention group and 58 partners from the control group.
Measure: Number (95% Confidence Interval); unit: percentage of casual male partners
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 110 | 58
percentage of casual male partners | 21.8 [15.1 to 30.4] | 10.3 [4.8 to 20.8]
Statistical Analysis 1: Comparison: Crowdsourced HIV PS Group vs Conventional HIV PS Group; Test type: Superiority; p = 0.07, Generalized linear regression

9. Secondary Outcome: Percentage of Presenting Partners Reporting Condom Use During the Last Anal Intercourse
Description: The percentage of presenting partners who completed the partner survey and reported condom use during the last anal intercourse
Time Frame: 3 months post enrollment
Population: Only 24 partners in the intervention group and 6 partners in the control group completed the partner survey that asked about their condom use during the last anal intercourse.
Measure: Number (95% Confidence Interval); unit: percentage of presenting partners
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
Number analyzed (Participants) | 24 | 6
percentage of presenting partners | 62.5 [42.7 to 78.8] | 33.3 [9.7 to 70.0]
Statistical Analysis 1: Comparison: Crowdsourced HIV PS Group vs Conventional HIV PS Group; Test type: Superiority; p = 0.11, Generalized linear regression

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed Consent through follow up, a total of approximately 3 months
Description: Adverse events are defined as an index reporting negative consequences after HIV disclosure to sexual partners, such as suffering violence.
Arm/Group | Crowdsourced HIV PS Group | Conventional HIV PS Group
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/40
Other Adverse Events (participants affected / at risk) | 1/81 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crowdsourced HIV PS Group (N=81) | Conventional HIV PS Group (N=40)
Negative consequences after HIV PS (Social circumstances) | 1 (1) | 0 (0) — One index in the intervention group reported suffering violence and getting divorced from his female partner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04971967/Prot_SAP_ICF_000.pdf